CLINICAL TRIAL: NCT05124535
Title: Population-based Age-stratified Seroepidemiological Investigation Protocol for Coronavirus 2019 (COVID-19) Infection in the Federation of Bosnia and Herzegovina
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute for Public Health of the Federation of Bosnia and Herzegovina (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2021-11-16; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Seroprevalence; Antibody; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Persons aged 18-29
- Persons aged 30-39
- Persons aged 40-65

SUMMARY:
This study is the second cross-sectional study conducted in the region. In the first cross sectional study, conducted in the winter of 2020, we aimed to estimate the seroprevalence of SARS-CoV-2 IgG antibodies among blood donors in Sarajevo Canton. We also assessed immune durability among seropositive participants after 6 months. In total, of 1015 blood donors aged 18-65 years in Sarajevo Canton between 2 November and 3 December 2020 were recruited and population-weighted seroprevalence in Sarajevo Canton was 19.2% (95% CI: 16.7-21.6%). The aim of this second cross-sectional study is to measure the seroprevalence SARS-CoV-2 antibodies and assess antibody kinetics in the blood donor population after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All individuals identified for recruitment into the investigation, resident of Canton Sarajevo between 18-65 years, irrespective of prior COVID-19 infection.

Exclusion Criteria:

* Refusal to give informed consent or to attend follow-up appointments; currently experiencing COVID-19 symptoms or in the last 14 days; and close contact with a confirmed case of COVID-19 within 14 days prior to donation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will be convenience sampling of blood donors aged between 18 and 65 years. All blood donors visiting the Institute for Transfusion Medicine of the Federation of Bosnia and Herzegovina for routine blood donation will be approached during the study period to participate in the study by the staff (medical doctors) of Institute for Transfusion Medicine of the Federation of Bosnia and Herzegovina at time of donation. Some blood donors will also be called by the staff of the Institute for Transfusion Medicine during the routine actions for donation of missing blood types, from an existing list maintained by staff at the Institute for Transfusion Medicine, and will be also invited to participate in the study by staff upon attendance at the blood clinic. Investigators will endeavor to ensure that the following three age groups can be reported: 18-29, 30-39, 40-65.
Sampling Method: Non-Probability Sample
Enrollment: 1152 (Estimated)
Dates: Start 2021-11-17 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence of SARS-CoV-2 IgG antibodies | November 2021-December 2021
  Crude seroprevalence among blood donors will be adjusted to age and sex distribution in cantonal population and to test sensitivity and specificity using Bayesian statistical modeling.

SECONDARY OUTCOMES:
Assess factors associated with seropositivity. | November 2021-December 2021
  Chi-squared test will be conducted on categorical variables.
Assess antibody response across types of immunity. | November 2021-December 2021
  Among those with positive anti-S antibodies, geometric mean titers will be compared across participants with natural immunity, vaccine-induced immunity, and hybrid of natural and vaccine-induced immunity.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Transfusion Medicine of the Federation of Bosnia and Herzegovina, Sarajevo, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided
If the data is shared by the implementing organization to WHO or any agency or institution providing support for data analysis, data shared will include only the study identification number and not any personally identifiable information.

REFERENCES:
- [Derived] Musa S, Catovic Baralija E, Ivey Sawin V, Nardone A, Palo M, Skocibusic S, Blazevic M, Cilovic Lagarija S, Ahmetovic-Karic G, Ljuca A, Dostovic-Halilovic S, Nedic R, Subissi L, Ibrahim R, Boshevska G, Bergeri I, Pebody R, Vaughan A. Evolution of seroprevalence to SARS-CoV-2 in blood donors in Sarajevo Canton, Federation of Bosnia and Herzegovina: Cross-sectional and longitudinal studies. Influenza Other Respir Viruses. 2023 Aug 22;17(8):e13182. doi: 10.1111/irv.13182. eCollection 2023 Aug. PMID 37621919